CLINICAL TRIAL: NCT00055679
Title: Phase III Randomized Study Of Adjuvant Fluourouracil, Epirubicin And Cyclophosphamide, In Women With Stage I Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Stage I Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACS05 UC-0140-0106; FRE-FNCLCC-PACS-05/0106; EU-20239
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 FEC (Active Comparator): 6 cycles of CYCLOPHOSPHAMIDE + EPIRUBICINE + 5-FLUOROURACILE
  Interventions: Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil
- 4 FEC (Experimental): 4 cycles of CYCLOPHOSPHAMIDE + EPIRUBICINE + 5-FLUOROURACILE
  Interventions: Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil

INTERVENTIONS:
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating early breast cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of different regimens of combination chemotherapy in treating women who have stage I breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of 4 vs 6 courses of adjuvant fluorouracil, epirubicin, and cyclophosphamide, in terms of 5-year survival, in women with stage I breast cancer.
* Compare the toxicity of these regimens in these patients.
* Determine the correlation of length of survival with biological factors in patients treated with these regimens.
* Determine biological factors significant for prognosis and prediction of survival of patients treated with these regimens.
* Determine the overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fluorouracil IV, epirubicin IV, and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive the same regimen as in arm I for up to 4 courses. After completion of chemotherapy, patients undergo radiotherapy 5 days a week for 6 weeks. Patients who are estrogen or progesterone receptor positive also receive oral tamoxifen daily for 5 years, beginning after completion of chemotherapy.

Patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 1,512 patients (756 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nonmetastatic, unilateral adenocarcinoma of the breast

  * Stage I
  * No clinically or radiologically suspicious metastases
  * No positive sentinel lymph nodes by immunohistochemistry for tumors less than 2 cm
  * No clinically proven positive axillary lymph nodes

    * Tumor cells found on immunohistochemistry only allowed
  * No clinically or radiologically contralateral suspicious lesions
* No deeply adherent disease
* No cutaneous invasion
* No inflammatory disease
* Complete surgical resection within the past 42 days

  * At least 8 lymph nodes removed
* Tumor at least 1 cm with no residual disease
* Presenting with at least 1 of the following factors of a poor prognosis:

  * Tumor greater than 2 cm
  * Hormone receptor negative tumor
  * Grade II or III
  * 35 years old or under
* Hormone receptor status:

  * Positive or negative

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Sex

* Female

Menopausal status

* Not specified

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST and ALT no greater than 1.25 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* No chronic hepatitis B
* No active hepatitis C

Renal

* Creatinine no greater than 1.25 times ULN

Pulmonary

* FEV normal

Other

* Not pregnant or nursing
* HIV negative
* No prior breast cancer or other malignancy
* No familial, social, or geographical reason that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No prior anticancer hormone therapy

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1512 (Actual)
Dates: Start 2002-08; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy, in terms of 5-year survival | 5 years from randomization

SECONDARY OUTCOMES:
Event free survival | 5 years from randomization
Toxicity | 5 years from randomization
Biological factors significant for prognosis and prediction of survival | 5 years from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kerbrat, MD, PhD, Study Chair — Centre Eugene Marquis
Locations (72):
- France (72):
  - Clinique Claude Bernard, Albi
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospital General Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Cote Basque, Bayonne
  - C.H.G. Beauvais, Beauvais
  - Centre Hospitalier General, Belfort
  - Institut Bergonie, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Hospitalier de Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier Jacques-Coeur, Bourges
  - CHU Hopital A. Morvan, Brest
  - Centre Hospitalier General, Brivé
  - Polyclinique Du Parc Centre Maurice Tubiana, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Regional de Chambery, Chambéry
  - Clinique Prive Paul d'Egine, Champigny-sur-Marne
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Clinique des Cedres, Cornebarrieu
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Draguignan, Draguignan
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Institut Prive de Cancerologie, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Hopital Andre Mignot, Le Chesnay
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Bretagne Sud, Lorient
  - Hopital Hotel Dieu, Lyon
  - Hopital de la Croix Rousse, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot, Lyon
  - Centre de Radiotherapie et Oncologie Saint-Faron, Mareuil-lès-Meaux
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier General Andre Boulloche, Montbéliard
  - Intercommunal Hospital, Montfermeil
  - Centre Azureen de Cancerologie, Mougins
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Clinique D'Occitanie, Muret
  - Centre Catherine de Sienne, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint-Herblain
  - Clinique Les Genets, Narbonne
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - C.H.G. De Pau, Pau
  - Clinique Saint - Pierre, Perpignan
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Centre Hospitalier de Cornouaille, Quimper
  - Centre Eugene Marquis, Rennes
  - CHG Roanne, Roanne
  - Centre Hospitalier de Rodez, Rodez
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Centre Medico-Chirurgical Foch, Suresnes
  - Polyclinique de L'Ormeau, Tarbes
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique Du Parc, Toulouse
  - Clinique du Chateau, Toulouse
  - Hopital J. Ducuing, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Kerbrat P, Desmoulins I, Roca L, Levy C, Lortholary A, Marre A, Delva R, Rios M, Viens P, Brain E, Serin D, Edel M, Debled M, Campone M, Mourret-Reynier MA, Bachelot T, Foucher-Goudier MJ, Asselain B, Lemonnier J, Martin AL, Roche H. Optimal duration of adjuvant chemotherapy for high-risk node-negative (N-) breast cancer patients: 6-year results of the prospective randomised multicentre phase III UNICANCER-PACS 05 trial (UCBG-0106). Eur J Cancer. 2017 Jul;79:166-175. doi: 10.1016/j.ejca.2017.03.004. Epub 2017 May 11. PMID 28501763